CLINICAL TRIAL: NCT01359735
Title: A Phase II Randomized, Open-label Study Investigating the Healing Effects of HP802-247 Versus Antibiotic Ointment in Mohs Micrographic Surgery Patients
Brief Title: Healing Effects of HP802-247 Versus Antibiotic Ointment in Mohs Micrographic Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 802-247-09-022
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Non-melanoma Skin Cancer
Keywords: Wound; non-melanoma skin cancer; Mohs micrographic surgery; Head or neck
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HP802-247 (Active Comparator): allogeneic, growth arrested keratinocytes and fibroblasts: final concentration of 5.0 M cells/mL with a ratio of 1:9 keratinocytes:fibroblasts, applied weekly
  Interventions: Biological: HP802-247
- Bacitracin Ointment (Active Comparator): bacitracin antibiotic ointment
  Interventions: Biological: Bacitracin Ointment

INTERVENTIONS:
Biological: HP802-247 — High dose HP 802-247, applied at each visit (Week 1-13) or until healed
  Arms: HP802-247
Biological: Bacitracin Ointment — One dose of Bacitracin ointment consists of 50 units/1 gram. This will be applied daily for 12 weeks (or until healed).
  Arms: Bacitracin Ointment

SUMMARY:
This study compares HP802-247 versus an antibiotic ointment for healing the wound after Mohs surgery.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Age ≥ 18 years and of either sex.
* Type I, II, or III skin as assessed by the Fitzpatrick Scale.
* Willing to comply with protocol instructions, including allowing all study assessments.
* Scheduled to have head or neck non-melanoma skin cancers removed by Mohs micrographic surgery with final wound size of 8 mm to 20 mm in diameter or with 8 mm to 20 mm long axis if not circular.
* Acceptable state of health and nutrition, in the opinion of the Investigator.

Exclusion Criteria:

* History of anaphylaxis, serum sickness, or erythema multiforme reaction to aprotinin, bovine serum albumin or bovine serum proteins, penicillin, streptomycin, or amphotericin B.
* Therapy with blood-thinning agents including aspirin within 14 days of the Baseline Visit (these may be resumed post-surgery).
* Subjects with platelet or coagulation disorders.
* Therapy with another investigational agent within thirty (30) days of Screening, or during the study.
* Current systemic therapy with cytotoxic drugs.
* Current therapy with chronic (> 10 days) oral corticosteroids.
* In the opinion of the Investigator the subject has a current life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint
Locations (1):
- Derm Research PLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a single US investigational site, between June 22, 2011and November 16, 2011
Pre-assignment Details: Subjects who met inclusion criteria returned for visit1 on the day of surgery and entered the study following. Subjects randomly assigned to HP802-247 or Bacitracin for post-surgical treatment, which lasted for up to 12 weeks or wound closure, which ever occurred first. Following completion of treatment subjects were followed for 4 weeks
Period: Overall Study
Arm/Group | HP802-247 | Bacitracin Ointment
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HP802-247 | Bacitracin Ointment | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (11.6) | 66.8 (10.7) | 70.4 (11)
Age, Customized [Number; unit: participants]
  50-69 yrs | 2 | 2 | 4
  70+ yrs | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Measure Was the Investigator's Global Assessment of Healing (IGAH).
Description: The IGAH is a four-point scale based on the following assessment scores: 0 = not effective, 1 = slightly effective, 2 = moderately effective, 3 = very effective. The descriptive statistics for both a continuous variable and a categorical variable were summarized for IGAH by treatment week and treatment endpoint. The Wilcoxon rank-sum test was used to test the difference in IGAH score between HP802-247 and bacitracin ointment for each treatment week and treatment endpoint. Since this was a small and exploratory study, the P-value of a 1-sided test was reported.
Time Frame: 13 weeks- The IGAH was measured at study Weeks 4 and 13
Population: The ITT population - all subjects who underwent MMS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HP802-247 | Bacitracin Ointment
Number analyzed (Participants) | 4 | 4
units on a scale
  Week 04 | 2.75 (0.5) | 2.25 (0.96)
  Week 13 | 3.00 (0) | 3.00 (0)
Statistical Analysis 1: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.263, Wilcoxon (Mann-Whitney) — Week 04
Statistical Analysis 2: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.500, Wilcoxon (Mann-Whitney) — Week 13

2. Secondary Outcome: The Number of Subjects With Complete Wound Closure at Each Evaluation Visit.
Description: Complete wound closure was assessed at each evaluation visit.
Time Frame: Over 12 weeks or until wound closure, which ever occurred first. Following completion of treatment subjects were followed for a further 4 weeks
Population: The ITT population - all subjects who underwent MMS. Fisher's exact test was used to examine the difference in proportion of subjects with complete wound closure at each of the corresponding time points between the two treatment groups, and the P-value of a 1-sided test was reported.
Measure: Number; unit: participants
Arm/Group | HP802-247 | Bacitracin Ointment
Number analyzed (Participants) | 4 | 4
participants
  Week 01 | 0 | 0
  Week 02 | 0 | 0
  Week 03 | 0 | 0
  Week 04 | 3 | 2
  Week 13 | 4 | 4
  Week 17/Exit | 4 | 4
Statistical Analysis 1: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.5, Fisher Exact — Over weeks 1 through 4 or Week 4?

3. Secondary Outcome: Time in Days to Wound Closure
Description: The Kaplan-Meier survival analysis was used to calculate the mean time in days to complete wound closure.
Time Frame: Over the 12 week treatment period
Population: The ITT population - all subjects who underwent MMS. The Log-rank test was used to test for an inter-group difference.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HP802-247 | Bacitracin Ointment
Number analyzed (Participants) | 4 | 4
Days | 24.8 (2.1) | 28.0 (3.5)
Statistical Analysis 1: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.0594, Log Rank

4. Secondary Outcome: Investigator Reported Signs and Symptoms
Description: Investigator reported signs and/or symptoms, based on the following 12 items, each scored as none (=0), mild (=1), moderate (=2), or severe (=3): Erythema, Erosion, Ulceration, Swelling, Scarring, Infection, Crusting, Necrosis, Peeling, Contact Dermatitis, Hyper/Hypopigmentation. Item scores were averaged.
Time Frame: At each evaluation visit: Weeks 3 and 12 post-surgery.
Population: The ITT population-all subjects who underwent MMS. Both total score and individual item score of the two signs and symptoms rating scales summarized descriptively at Weeks 4, 7, and 13 as well as at the treatment endpoint and compared using a two-sample t-test. the P-value of a 1-sided test was reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HP802-247 | Bacitracin Ointment
Number analyzed (Participants) | 4 | 4
units on a scale
  3 Weeks Post Surgery | 1.75 (0.96) | 3 (1.83)
  12 Weeks Post Surgery | 1.00 (0.82) | 1.00 (0.82)
Statistical Analysis 1: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.1354, t-test, 1 sided — 3 Weeks
Statistical Analysis 2: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.5000, t-test, 1 sided — 12 Weeks

5. Secondary Outcome: Subject Reported Signs and Symptoms
Description: Subjects reported signs or symptoms, based on the following 6 items, each scored as none (=0), mild (=1), moderate (=2), or severe (=3): irritation, itchiness, burning, tenderness, pain, and stinging. Item scores were averaged.
Time Frame: At each evaluation visit: Weeks 3, and 12 post-surgery.
Population: The ITT population - all subjects who underwent MMS. Both the total score and individual item score of the two signs and symptoms rating scales were summarized descriptively at Weeks 4, 7, and 13 as well as at the treatment endpoint and compared using a two-sample t-test, and the P-value of a 1-sided test was reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HP802-247 | Bacitracin Ointment
Number analyzed (Participants) | 4 | 4
units on a scale
  Week 3 Post-surgery | 0 (0) | 0.75 (0.96)
  Week 12 Post-surgery | 0.25 (0.50) | 0 (0)
Statistical Analysis 1: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.0841, t-test, 1 sided — Week 3 Post-surgery
Statistical Analysis 2: Comparison: HP802-247 vs Bacitracin Ointment; Test type: Superiority or Other; p = 0.1780, t-test, 1 sided — Week 12 Post-surgery

ADVERSE EVENTS:
Time Frame: Safety reporting occurred over the eight weeks of the study.
Description: All subjects randomized to treatment were questioned about adverse events and were included in the number of participants assessed for safety. The first assessments at each visit were about changes in general health and concomitant medications and the occurrence of adverse events.
Arm/Group | HP802-247 | Bacitracin Ointment
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 (N=4) | Bacitracin Ointment (N=4)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less